CLINICAL TRIAL: NCT03811509
Title: Study for Improving Life Quality in Breast Cancer Women Treated With Aromatase Inhibitors: Cohort B-ABLE
Brief Title: Breast Cancer Women on Aromatase Inhibitors Treatment
Acronym: B-ABLE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4604010730
Record Dates: First submitted 2018-12-17; First posted 2019-01-22 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2018-08

CONDITIONS: Osteoporosis; Osteoporosis Fracture; Arthralgia Generalized
Keywords: osteoporosis; aromatase inhibitors; breast cancer; microindentation; arthralgia; musculoskeletal pain
MeSH Terms: conditions — Osteoporosis; Osteoporotic Fractures; Breast Neoplasms; Arthralgia; Musculoskeletal Pain | interventions — Diphosphonates; Denosumab

STUDY DESIGN:
Intervention Model Description: All patents receive aromatase inhibitors Patients without osteoporosis receive only calcium and vitamin D Patients with osteoporosis receive antiresorptive treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI with osteoporosis (Active Comparator): Patients with osteoporosis receive intervention with antiresorptive treatment, bisphosphonates or denosumab . All patients receive calcium and Vit D supplements All patients receive by protocol aromatase inhibitors for breast cancer treatment, letrozole, exemestane for 5 o 10 years.
  Interventions: Drug: bisphosphonate
- AI without osteoporosis (No Intervention): All patients receive calcium and Vit D supplements All patients receive by protocol aromatase inhibitors for breast cancer treatment, letrozole, exemestane for 5 o 10 years.

INTERVENTIONS:
Drug: bisphosphonate — antiresorptives
  Other Names: denosumab
  Arms: AI with osteoporosis

SUMMARY:
The main objective of the study is to improve the life quality of women treated with AI. Cohort B-ABLE is designed to evaluate musculoskeletal events derived of using AI in breast cancer women. The project objectives are the analysis of the AI deleterious effect on bone microarchitecture and early determination of the risk of fragility fracture with dual energy x-ray absorptiometry (DEXA), lumbar spine Rx, Trabecular Bone Score (TBS) and microindentation. Determination of physiological causes of the AI-related arthralgia by analyzing joint degradation markers, steroid hormone levels remaining in blood and functional magnetic resonance, before and after three months of AI treatment

DETAILED DESCRIPTION:
Postmenopausal women with breast cancer treated with aromatase inhibitors (AI) have a higher incidence of osteoporosis, fractures and other musculoskeletal symptoms, particularly pain and stiffness. B-ABLE is a clinical, prospective cohort study carried out in both Breast Cancer and Bone Metabolism Units of the Hospital del Mar in Barcelona. Currently, 780 postmenopausal Caucasian women with early breast cancer and candidates for adjuvant AI treatment were included and predicted to reach more than 1000 patients. The main objective of the study is to improve the life quality of women treated with AI. Cohort B-ABLE is designed to evaluate musculoskeletal events derived of using AI in breast cancer women. The project objectives are the analysis of the AI deleterious effect on bone microarchitecture and early determination of the risk of fragility fracture with DEXA, lumbar spine Rx, TBS and microindentation. Determination of physiological causes of the AI-related arthralgia by analyzing joint degradation markers, steroid hormone levels remaining in blood and functional magnetic resonance, before and after three months of AI treatment. The study results will help to decide the most appropriate treatment for each patient in order to minimize AI-related side effects and hence avoid discontinuation of adjuvant therapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with early breast cancer estrogen receptor with aromatase inhibitors treatment

Exclusion Criteria:

* Previous treatment with antiresorptive treatment for osteoporosis secondary osteoporosis, as corticosteroids, Hyperparathyroidism, Kidney Chronic disease, previous treatment with aromatase inhibitors Diabetes mellitus type 1 Fibromyalgia

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
bone mass measured by dual energy x-ray absorptiometry (DEXA) densitometry | change from baseline, 12 months, 24 months, 36 months, 48 months 60 months and 1 year after completion of aromatase treatment
  bone mas normal, osteopenia or osteoporosis related with WHO definition of osteoporosis and Trabecular Bone Score: normal, mild degratation and high degradation
Fragility fractures assessed by xRay | incidence of new fractures at 12 months, 24 months, 36 months, 48 months 60 months of aromatase treatment
  vertebral and non vertebral fractures, hip fractures
Bone Mineral Strength (BMSi) | change from baseline, 12 months, and 60 months of aromatase treatment
  bone microindentation
Arthralgia | change from baseline, 12 months, 24 months, 36 months, 48 months 60 months and 1 year after completion of aromatase treatment
  joint pain measured by analogic visual scale range 0= no pain 10= worse pain

SECONDARY OUTCOMES:
bone turnover markers | change from baseline, 12 months, 24 months, 36 months, 48 months 60 months and 1 year after completion of aromatase treatment
  C-telopeptide (Ctx), Procollagen type 1 amino-terminal propeptide (P1NP) Bone Alkaline Phosphatase (AP)
cartilage degradation markers | change from baseline and 12 months of aromatase treatment
  C-telopeptide II, Procollagen type 2 amino-terminal propeptide (P2NP)

CONTACTS AND LOCATIONS:
Locations (1):
- Xavier Nogues, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Publication in Oncology , Endocrinology and bone metabolism journals
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available in the next year and every time we have outcomes available
Access Criteria: By asking CEIC Parc de Salut Mar

REFERENCES:
- [Background] Servitja S, Nogues X, Prieto-Alhambra D, Martinez-Garcia M, Garrigos L, Pena MJ, de Ramon M, Diez-Perez A, Albanell J, Tusquets I. Bone health in a prospective cohort of postmenopausal women receiving aromatase inhibitors for early breast cancer. Breast. 2012 Feb;21(1):95-101. doi: 10.1016/j.breast.2011.09.001. Epub 2011 Sep 15. PMID 21924904
- [Background] Nogues X, Servitja S, Pena MJ, Prieto-Alhambra D, Nadal R, Mellibovsky L, Albanell J, Diez-Perez A, Tusquets I. Vitamin D deficiency and bone mineral density in postmenopausal women receiving aromatase inhibitors for early breast cancer. Maturitas. 2010 Jul;66(3):291-7. doi: 10.1016/j.maturitas.2010.03.012. Epub 2010 Apr 15. PMID 20399042
- [Result] Servitja S, Martos T, Rodriguez Sanz M, Garcia-Giralt N, Prieto-Alhambra D, Garrigos L, Nogues X, Tusquets I. Skeletal adverse effects with aromatase inhibitors in early breast cancer: evidence to date and clinical guidance. Ther Adv Med Oncol. 2015 Sep;7(5):291-6. doi: 10.1177/1758834015598536. PMID 26327926
- [Derived] Pineda-Moncusi M, Servitja S, Tusquets I, Diez-Perez A, Rial A, Cos ML, Campodarve I, Rodriguez-Morera J, Garcia-Giralt N, Nogues X. Assessment of early therapy discontinuation and health-related quality of life in breast cancer patients treated with aromatase inhibitors: B-ABLE cohort study. Breast Cancer Res Treat. 2019 Aug;177(1):53-60. doi: 10.1007/s10549-019-05289-7. Epub 2019 May 24. PMID 31127467